CLINICAL TRIAL: NCT01822314
Title: Neoadjuvant Chemotherapy With Nab-paclitaxel in Women With HER2-negative High-risk Breast Cancer " ETNA (Evaluating Treatment With Neoadjuvant Abraxane)
Brief Title: Neoadjuvant Chemotherapy With Nab-paclitaxel in Women With HER2-negative High-risk Breast Cancer
Acronym: ETNA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fondazione Michelangelo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FM-12-B01; 2012-003481-41 (EudraCT Number)
Record Dates: First submitted 2013-03-25; First posted 2013-04-02 (Estimated); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Breast Cancer
Keywords: breast; cancer; unilateral; non metastatic; HER2 negative
MeSH Terms: conditions — Breast Neoplasms; Neoplasms | interventions — Albumin-Bound Paclitaxel; 130-nm albumin-bound paclitaxel; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Paclitaxel (Active Comparator): Paclitaxel will be given on week 1, 2 and 3 followed by 1 week rest and will be repeated for 4 cycles.
  AC or EC or FEC will then be given on day 1 every 3 weeks for 4 cycles
  Interventions: Drug: Paclitaxel
- Abraxane (Experimental): Abraxane will be given at the dosage of 125 mg/m2 on week 1, 2 and 3 followed by 1 week rest and will be repeated for 4 cycles.
  AC or EC or FEC will then be given on day 1 every 3 weeks for 4 cycles
  Interventions: Drug: Abraxane

INTERVENTIONS:
Drug: Abraxane — Abraxane at the dosage of 125 mg/m2 will be delivered over 30 minutes on week 1, 2 and 3 followed by 1 week rest. week rest and will be repeated for 4 cycles followed by AC or EC (adriamycin or epirubicin and cyclophosphamide) on day 1 every 3 weeks for 4 cycles or FEC (fluorouracil, epirubicin, and cyclophosphamide) on day 1 every three weeks for 4 cycles
  Other Names: Nab-paclitaxel
  Arms: Abraxane
Drug: Paclitaxel — Paclitaxel at the dosage of 90 mg/m2 diluted in 250 mL of water for injection (WFI) over 1 hour given week 1, 2 and 3 followed by 1 week rest and will be repeated for 4 cycles followed by AC or EC (adriamycin or epirubicin and cyclophosphamide) on day 1 every 3 weeks for 4 cycles or FEC (fluorouracil, epirubicin, and cyclophosphamide) on day 1 every three weeks for 4 cycles
  Other Names: No specific brand name
  Arms: Paclitaxel

SUMMARY:
The purpose of this study is to assess the efficacy of neoadjuvant weekly nab-paclitaxel followed by Adriamycin, Cyclophosphamide (AC) or Epirubicin, Cyclophosphamide (EC) or Fluorouracil,Epirubicin,Cyclophosphamide (FEC)compared with neoadjuvant weekly solvent-based paclitaxel followed by AC or EC or FEC in terms of rate of pathological complete remissions at surgery.

DETAILED DESCRIPTION:
In this study, eligible and consenting patients will be randomized to receive either 4 cycles of weekly abraxane (nab-paclitaxel) followed by 4 cycles of an anthracycline-containing regimen or 4 cycles of weekly paclitaxel followed by 4 cycles of an anthracycline-containing regimen.The anthracycline regimen (AC, EC or FEC) will be chosen by the investigator at the participating sites.

Before randomization patients will be stratified according to Disease stage [operable (tumor stage: T2N0-1; T3N0) and locally advanced (T3N1;T4, any N2-3)] and Tumor subtype [luminal B intermediate (HER2 negative, ER or PGR positive, Ki67 from 14% to 20%) vs luminal B high (HER2 negative, ER or PGR positive, Ki67 >20%) vs triple negative tumors (HER2 negative, ER negative and PgR negative, Ki67 any value)]. Tumor subtype will be confirmed at two selected referral laboratories.

Neoadjuvant chemotherapy will be followed by definite surgery and irradiation as per international and local guidelines.

During neoadjuvant chemotherapy patients will be assessed for safety and efficacy as detailed in the protocol.

After definite surgery patients will be followed for approximately 10 years according to local procedures

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged 18 years or older
* Histologically confirmed invasive unilateral breast cancer
* HER2-negative disease
* Known hormone receptor status (estrogen receptor [ER], progesterone receptor [PgR]), tumor grade and, if institutional standard permits, known Ki67 value
* Available paraffin-embedded tumor block taken at diagnostic biopsy for central confirmation of HER2 eligibility, hormone receptor status, Ki67 value and biomarker evaluation is mandatory
* One of the following clinical stages:
* T2, T3, T4 disease, triple negative (HER2, ER, PgR)
* T2, T3, T4 disease, ER or PgR positive and moderately differentiated or poorly differentiated tumor grade (G II-III)
* ECOG performance status 0 or 1
* Written informed consent to participate in the trial (approved by the Institutional Review Board [IRB]/ Independent Ethics Committee [IEC]) obtained prior to any study specific screening procedures
* Willing and able to comply with the protocol

Exclusion Criteria:

* Synchronous contralateral breast cancer or presence of metastatic disease (M1). Exception: contralateral insitu ductal cancer
* Surgical axillary staging procedure prior to study entry. Exceptions: 1) Fine needle aspiration (FNA) of an axillary node is permitted for any patient, and 2) although not recommended, a pre-neoadjuvant therapy sentinel lymph node biopsy for patients with clinically negative axillary nodes is permitted
* Pregnant or lactating women.
* Women with childbearing potential unless (1) surgically sterile or (2) using adequate measures of contraception, for example abstinence, an intra-uterine device, or double barrier method of contraception
* Treatment including radiation therapy, chemotherapy, biotherapy, and/or hormonal therapy for the currently diagnosed breast cancer prior to study entry
* Previous investigational treatment for any condition within 4 weeks of randomization date
* Patients on therapy with a strong CYP3A4 inhibitor and on therapy with Warfarin (Coumadin)
* Previous or concomitant malignancy of any other type that could affect compliance with the protocol or interpretation of results. Patients with curatively treated basal cell carcinoma of the skin or in situ cervix cancer are generally eligible.
* Pre-existing motor or sensory neuropathy of grade > 1 for any reason
* Patients with a history of hypersensitivity due to drugs containing polyoxyethylene castor oil (Cremophor EL) (e.g., ciclosporin), or hardened castor oil (e.g., vitamin preparations for injection, etc.)
* Other serious illness or medical condition including: history of documented congestive cardiac failure; angina pectoris requiring anti-anginal medication; evidence of transmural infarction on ECG; poorly controlled hypertension (e.g. systolic >180 mm Hg or diastolic >100 mm Hg; however, patients with hypertension which is well controlled on medication are eligible); clinically significant valvular heart disease; high-risk uncontrolled arrhythmias
* Patients with a history of uncontrolled seizures, central nervous system disorders or psychiatric disability judged by the investigator to be clinically significant and precluding informed consent or adversely affecting compliance with study drugs
* Serious uncontrolled infections (bacterial or viral) or poorly controlled diabetes mellitus
* Hematology and biochemistry tests within normla limits
* Baseline left ventricular ejection fraction (LVEF) < 50% by echocardiography or multi-gated scintigraphic scan (MUGA)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 632 (Actual)
Dates: Start 2013-04; Primary Completion 2016-09 (Actual); Study Completion 2023-03 (Actual)

PRIMARY OUTCOMES:
pathologic Complete Response (pCR) | At the time of surgery: 40 months after the randomization of the first patient
  To compare the rate of pathologic Complete Response (pCR, absence of invasive disease in breast and nodes (ypT0/ypTis, ypN0)) for abraxane (Abraxane®, abraxane) vs paclitaxel.

SECONDARY OUTCOMES:
clinical Overall Response (cOR) | At the time of surgery: 40 months after the randomization of the first patient
  To compare the rate of clinical overall response (cOR) after the first 4 cycles of abraxane vs paclitaxel and to compare the rate of cOR after the entire preoperative chemotherapy (i.e. before surgery) in the study arms of abraxane vs paclitaxel
Event Free Survival (EFS) | 5 years after the first patient in and 10 years after randomization of last patient in
  To compare the Event Free Survival (EFS, i.e. disease progression while on primary therapy or disease recurrence after surgery) in the study arms of abraxane vs paclitaxel
Distant Event Free Survival (DEFS) | 5 years after the first patient in and 10 years after randomization of last patient in
  The distant event free survival (DEFS) is defined as the time from randomization to the first date of distant metastasis while on primary therapy or distant recurrence after surgery or death due to any cause. Patients who terminate the study without evidence of any of the above events will be censored at the date of their last follow-up tumor assessment
Local Event Free Survival | 5 years after the first patient in and 10 years after randomization of last patient in
  The local event free survival (LEFS) is defined as the time from randomization to the first date of local progression while on primary therapy or local recurrence after surgery. Rules for censoring and methods of analysis will be the same as defined for EFS
Regional Event Free Survival | 5 years after the first patient in and 10 years after randomization of last patient in
  The regional event free survival (REFS) is defined as the time from randomization to the first date of regional progression while on primary therapy or regional recurrence after surgery. Rules for censoring and methods of analysis will be the same as defined for EFS.
Overall Survival (OS) | 13 years from the date of first patient in
  The overall survival (OS) is defined as the time from randomization to the date of death. Patients alive at the end of study will be censored at their last contact date.
Safety and Tolerability | Each participant will be followed for the duration of treatment period, approximately 9 months
  Patients will be assessed for adverse events by clinical examination, questioning for symptoms of toxicity, laboratory assessments, vital signs, ECG and LVEF.
  Neurological toxicity and other toxicities will be assessed throughout the study according the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Event (CTCAE) Version 4.0.

CONTACTS AND LOCATIONS:
Overall Officials: Luca Gianni, MD, Study Chair — San Raffaele Hospital, Milan
Locations (66):
- Australia (7):
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Peter McCallum Cancer Centre, East Melbourne, Victoria
  - Peter MacCallum Cancer Centre Department of Surgical Oncology, East Melbourne, Victoria
  - Eastern Health Breast Cancer Research - Maroondah Breast Clinic, Ringwood East, Victoria
  - Eastern Health Breast Cancer Research Maroondah Breast Clinic, Ringwood East, Victoria
  - Mount Hospital - Breast Clinical Trials Unit, Perth, Western Australia
  - Royal Perth Hospital, Perth, Western Australia
- Germany (12):
  - Klinikum Augsburg International Patient Service, Augsburg
  - Frauenarzt-Zentrum-Zehlendorf, Berlin
  - Augusta-Kranken-Anstalt gGmbH Klinik für Hämatologie, Onkologie & Palliativmedizin, Bochum
  - St.Elisabeth-Krankenhaus Brustzentrum, Cologne
  - Universitätsklinikum Erlangen - Frauenklinik - Poliklinik, Erlangen
  - Agaplesion Markus Hospital - Frankfurt, Frankfurt
  - Bethanien-Krankenhaus Onkologisches Zentrum, Frankfurt
  - Mammazentrum - Hamburg am Krankenhaus Jerusalem, Hamburg
  - Gynäkologisch-Onkologische Praxis, Hanover
  - Interdisciplinary Oncology Center, Munich
  - Praxis Gynäkologie Arabella, Munich
  - Onkologische Schwerpunktpraxis, Speyer
- Italy (15):
  - Cliniche Gavazzeni - Humanitas Gavazzeni, Bergamo, BG
  - Policlinico Sant'Orsola Malpighi, Bologna, BO
  - Azienda Ospedaliero-Universitaria di Ferrara - Arcispedale Sant'Anna, Cona, Ferrara
  - IST San Martino, Genova, GE
  - A.O. San Gerardo, Monza, MB
  - A.O. Ospedale Civile di Legnano, Legnano, MI
  - Ospedale San Raffaele, Milan, MI
  - Fondazione IRCCS Istituto nazionale dei tumori, Milan, MI
  - A.O. Ospedale Luigi Sacco, Milan, MI
  - A.O. Ospedale Niguarda Ca' Granda, Milan, MI
  - ULSS 15 Alta Padovana, Camposampiero, PD
  - Fondazione IRCCS Policlinico San Matteo, Pavia, PV
  - Arcispedale Santa Maria Nuova, Reggio Emilia, RE
  - Ospedale Santa Maria della Misericordia, Udine, UD
  - Azienda ULSS 6 di Vicenza, Vicenza, VI
- NN Petrov Research Institute of Oncology, Saint Petersburg, Russia
- National Cancer Centre Singapore, Singapore, Singapore
- Spain (30):
  - Hospital Clinico Lozano Blesa, Zaragoza, Aragon
  - Miguel Servet University Hospital, Zaragoza, Aragon
  - Hospital Son Llàtzer Palma de Mallorca, Palma de Mallorca, Balearic Islands
  - Corporacio Sanitaria Parc Tauli, Sabadell, Barcelona
  - Consorci Sanitari de Terrassa, Terrassa, Barcelona
  - Hospital Universitario Fundacion Alcorcón, Alcorcón, Madrid
  - Hospital Universitario de Canarias, San Cristóbal de La Laguna, Tenerife
  - Centro Oncologico de Galicia, A Coruña
  - Hospital Teresa Herrera (Chuac), A Coruña
  - Hospital General Universitario de Alicante, Alicante
  - Hospital Nuestra Señora de Sonsoles, Ávila
  - Institut d'Investigació en Ciències de la Salut Germans Trias i Pujol, Badalona
  - Hospital del Mar, Barcelona
  - Hospital Clinic i Provencial, Barcelona
  - Hospital San Pedro de Alcantara, Cáceres
  - Hospital Universitario Reina Sofía, Córdoba
  - Onkologikoa, Donostia / San Sebastian
  - Complejo Hospitalario de Jaen, Jaén
  - Hospital Universitari Arnau de Vilanove de Lleida, Lleida
  - Gregorio Maraňón Hospital, Madrid
  - Hospital La Paz, Madrid
  - MD Anderson Cancer Center Madrid, Madrid
  - J.M. Morales Meseguer, Universitary Hospital Marques in los Velez, Murcia
  - Hospital Clinico Universitario de Salamanca, Salamanca
  - Hospital Universitario Donostia, San Sebastián
  - Hospital Virgen del Rocio, Seville
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Virgen de la Salud, Toledo
  - Instituto Valenciano Oncologia, Valencia
  - Hospital Clinico Universita Valencia, Valencia

REFERENCES:
- [Derived] Gianni L, Mansutti M, Anton A, Calvo L, Bisagni G, Bermejo B, Semiglazov V, Thill M, Chacon JI, Chan A, Morales S, Alvarez I, Plazaola A, Zambetti M, Redfern AD, Dittrich C, Dent RA, Magazzu D, De Fato R, Valagussa P, Tusquets I. Comparing Neoadjuvant Nab-paclitaxel vs Paclitaxel Both Followed by Anthracycline Regimens in Women With ERBB2/HER2-Negative Breast Cancer-The Evaluating Treatment With Neoadjuvant Abraxane (ETNA) Trial: A Randomized Phase 3 Clinical Trial. JAMA Oncol. 2018 Mar 1;4(3):302-308. doi: 10.1001/jamaoncol.2017.4612. PMID 29327055